CLINICAL TRIAL: NCT01085565
Title: Phase II Study to Evaluate the Safety and Effectiveness of ExAblate MR Guided Focused Ultrasound Surgery in the Treatment of Pain Resulting From Metastatic Bone Tumors With the ExAblate 2100 Conformal Bone System
Brief Title: Focused Ultrasound Surgery in the Treatment of Pain Resulting From Metastatic Bone Tumors With the ExAblate 2100 Conformal Bone System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM011
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Bone Cancer; Bone Metastases; Pain
Keywords: Bone cancer; Bone Metastases; pain palliation; metastasis; breast cancer; lung cancer; prostate cancer; cancer related pain; tumors
MeSH Terms: conditions — Bone Neoplasms; Pain; Neoplasm Metastasis; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Cancer Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exablate treatment (Experimental)
  Interventions: Device: ExAblate 2100

INTERVENTIONS:
Device: ExAblate 2100 — Conformal Bone System

SUMMARY:
The goal of this prospective, non-randomized, single-arm, phase 2 study is to evaluate the safety and effectiveness of this treatment using this ExAblate conformal system in the treatment of pain resulting from metastatic bone tumors Up to Fifty (50) patients will be recruited in this feasibility study. The treated patients will be followed for 3-Months post their last treatment, patients with the standard contraindications to MRI examination, such as implanted metal devices (pacemakers, etc.), will be excluded.

DETAILED DESCRIPTION:
Bone is the third most common organ involved by metastatic disease behind lung and liver [6]. In breast cancer, bone is the second most common site of metastatic spread, and 90% of patients dying of breast cancer have bone metastasis. Breast and prostate cancer metastasize to bone most frequently, which reflects the high incidence of both these tumors, as well as their prolonged clinical courses. Post-cancer survival has increased with improvement in early detection and treatments. As a consequence, the number of patients developing metastatic bone disease during their lifetime has also increased.

Current treatments for patients with bone metastases are primarily palliative and include localized therapies (radiation and surgery), systemic therapies (chemotherapy, hormonal therapy, radiopharmaceutical, and bisphosphonates although the primary goal of the use of these therapies are often to address the disease itself), and analgesics (opioids and non-steroidal anti-inflammatory drugs). Recently, radiofrequency ablation has been tested as a treatment option for bone metastases [8]. Currently, an off label use of Cryoablation techniques are being tested as another alternative for bone Mets palliation. The main goals of these treatments are improvement of quality of life and functional level. These goals can be further described:

1. Pain relief
2. Preservation and restoration of function
3. Local tumor control
4. Skeletal stabilization

Treatment with external beam radiation therapy (EBRT) is the standard of care for patients with localized bone pain, and results in the palliation of pain for many of these patients. Twenty to 30% of patients treated with radiation therapy do not experience pain relief [9-13]. Re-treatment rates are generally reported in the range of 10-25%. Many patients with relapsed pain or poor response to initial radiation may be lost to follow up or may not be referred back to oncologists for consideration of re-radiation. In addition to relapse and re-treatment, there is an increased risk of pathologic fracture in the peri-radiation period. The fracture rate reported in radiation studies is generally in the range of 1% to 8%. The hyperemic response weakens the adjacent bone and increases the risk of spontaneous fracture. Furthermore, patients who have recurrent pain at a site previously irradiated may not be eligible for further radiation therapy secondary to limitations in normal tissue tolerance. Hesitation on the part of physicians to use a larger dose may be related to increased long-term toxicity. Larger radiation dose produces a greater risk of complications such as fibrosis of normal soft tissue, which can cause a decrement in the quality of life in cases of life expectancy longer than 6 months. There may also be a greater incidence of acute side effects of nausea and vomiting if the treatment field includes the stomach. The percent of patients experiencing vomiting following EBRT ranges from about 5% to 30%.

A palliative treatment for painful bone metastases that is non-invasive, without long-term toxicity and having minimal complications would be a useful tool for treating physicians and also a beneficial option for patients suffering from painful bone metastases. Results of preliminary studies indicate that ExAblate treatment of painful bone metastases may be a beneficial treatment option [14, 15]. The ExAblate system is a non-invasive thermal ablation device used in the coagulation of various types of soft tissue. The ExAblate system has the potential to achieve the first three of the four previously mentioned goals in the treatment of bone tumors; namely pain relief, preservation and restoration of functional levels and local tumor control [11]. The ExAblate system used in the present study is a technological advance over the ExAblate 2000 fixed transducer system in terms of flexibility of use and reduction of positioning related pain to the patients. The ExAblate system used in this study conforms to the patient's body shape at the location of the bone mets location

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 and older
2. Patients who are able and willing to give consent and able to attend all study visits
3. Patients who are suffering from symptoms of bone metastases
4. Targeted tumor(s) are ExAblate device accessible and are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5)
5. Patient with NRS (0-10 scale) pain score ≥ 4 at the targeted tumors irrespective of medication.
6. Patient who's targeted tumors are on bone and bone-lesion interface is more than 1cm from the skin, major nerve or hollow viscera.
7. Targeted tumors clearly visible by non-contrast MRI, and ExAblate MRgFUS device accessible
8. Able to communicate sensations during the ExAblate MRgFUS treatment

Exclusion Criteria:

1. Patients who either:

   * Need surgical stabilization of the affected weight bearing bony structure OR
   * Targeted tumor is at an impending fracture site of the weigh bearing bone. OR
   * Patients with surgical stabilization of tumor site with metallic hardware
2. Target tumors-bone interface is less then 1cm from nerve bundles, bowels, skin or bladder.
3. Targeted (most painful) tumors:

   * NOT visible by non-contrast MRI, OR
   * NOT accessible to ExAblate device
4. Targeted tumor is in the skull
5. Patients on dialysis
6. Patients with life expectancy < 6-Months
7. Patients with an acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.
8. Subjects with Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication
   * Patients with documented myocardial infarction less than 40 days prior to protocol enrolment
   * Subjects with Severe Congestive Heart Failure, NYHA class 4.
   * Patients on anti-arrhythmic drugs or with uncontrolled and/or untreated arrhythmia status
9. Severe cerebrovascular disease (CVA within last 6 months)
10. Severe hypertension (diastolic BP > 100 on medication)
11. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
12. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
13. Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
14. KPS Score < 60 (See "Definitions" below)
15. Patients unable to communicate with the investigator and staff.
16. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.)
17. Are participating or have participated in another clinical trial for the palliation of their targeted bone metastasis tumors in the last 30 days
18. Patients receiving new chemotherapy regime or radiation to the targeted lesion (s) within the last two weeks
19. Patients with persistent undistinguishable pain (pain source unidentifiable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months post treatment
  Evaluate incidence and severity of adverse events associated with ExAblate MRgFUS ExAblate Conformal system used in the palliation of pain due to metastatic bone tumors

SECONDARY OUTCOMES:
Efficacy | 3 months post treatment
  Level of pain relief (measured by Pain Scale)
Effectiveness | 3 months post treatment
  Decrease in analgesics/opiate
Effectiveness | 3 months post treatment
  Improved quality of life (measured by questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba MC, Ramat Gan, Israel

REFERENCES:
- See also: Sponsor's website — http://www.insightec.com